CLINICAL TRIAL: NCT00998387
Title: Translation and Validation of the Korean Version of Confusion Assessment Method for the Intensive Care Unit
Brief Title: Validation of the Korean Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sang Min Lee M.D, Seoul National University Hospital
Other Study IDs: 0803-058-239
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- medical ICU: admitted to medical ICU at Seoul National University Hospital longer than 24 hours

SUMMARY:
The purpose of this study is to translate and validate the CAM-ICU for use in the Korean ICU setting.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* admitted to medical ICU at Seoul National University Hospital longer than 24 hours

Exclusion Criteria:

* comatose or moribund state throughout the study period
* preexisting neurologic problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to medical ICU at Seoul National University Hospital longer than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Interrater reliability of Korean CAM-ICU | after completion of study
Sensitivity of Korean CAM-ICU for diagnosing ICU delirium | after completion of study
Specificity of Korean CAM-ICU for diagnosing ICU delirium | after completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea